CLINICAL TRIAL: NCT03840265
Title: Evaluation of Cerebrovascular Events in Patients With Occlusive Carotid Artery Disorders Based on Morphological and Hemodynamical Features
Brief Title: Evaluation of Cerebrovascular Events in Patients With Occlusive Carotid Artery Disorders
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Semmelweis University Heart and Vascular Center (Other)
Collaborators: National Research, Development and Innovation Office (Unknown)
Responsible Party: Principal Investigator, Prof. Dr. Sótonyi Péter, MD, PhD, Head of Vascular Surgery Department of Semmelweis University, Semmelweis University Heart and Vascular Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: SemmelweisUHVC
Record Dates: First submitted 2019-02-12; First posted 2019-02-15 (Actual); Last update posted 2020-03-20 (Actual); Status verified 2020-03

CONDITIONS: Carotid Stenosis; Carotid Artery Plaque; Cerebrovascular Embolism and Thrombosis
MeSH Terms: conditions — Carotid Stenosis; Intracranial Embolism and Thrombosis | interventions — Endarterectomy, Carotid; Ultrasonography, Doppler, Transcranial

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Carotid endarterectomy (Other): All patients in this study will undergo carotid endarterectomy procedure
  Interventions: Procedure: carotid endarterectomy

INTERVENTIONS:
Procedure: carotid endarterectomy — In this project the following parameters will be assessed both in asymptomatic and symptomatic patients underwent carotid endarterectomy: 1) hemodynamic modeling of effect of the supraaortic arteries anatomic variations and pathologies 2, preoperative stroke risk prediction based on comparative analysis of CTA results of plaque morphology and ultrasound-based plaque elastography analysis, 3) cerebral flow measurement by transcranial Doppler sonography(TCD), 4) presence recent of silent brain ischemia on DWI-MRI, 5) OCT angiography could be a useful non-invasive method for evaluation of the outcome of carotid interventions
  Other Names: Cranial MR; Transcranial Doppler Ultrasound; Optical coherence tomography angiography; Carotid CT angiography

SUMMARY:
As of today, no suitable multiparametric predictive method is available to properly estimate stroke risk in patients with carotid artery stenosis. Carotid artery stenosis is one of the proven risk factors of stroke incidence, but the indication of its intervention is merely the grade of stenosis itself. The current international guidelines suggest intervention for asymptomatic patients only with potentially high risk plaques but pharmacological treatment is advised to low risk patients. Unfortunately there is no proven and widely accepted system to distinguish these two categories of patients with carotid artery stenosis.

In this project the following parameters will be assessed both in asymptomatic and symptomatic patients: 1, preoperative stroke risk prediction based on comparative analysis of CT angiography (CTA) results of plaque morphology and ultrasound (US) based plaque elastography analysis, 2) intracranial bloodflow will be measured by transcranial Doppler sonography(TCD), 3) presence recent of silent brain ischemia on diffusion weighted imaging (DWI) MR (magnetic resonance), 4) retinal perfusion measurement by optical coherence tomography angiography (OCT). The investigators aim to establish a clinically meaningful and more accurate (than stenosis grade) stroke risk prediction algorithm for asymptomatic carotid stenosis patients based on these parameters.

DETAILED DESCRIPTION:
Stroke is one of the leading causes of mortality in Hungary. While stroke mortality is 8-10/100.000 in the population under 50 years of age in Western European countries, the mortality is 40/100.000 in women and 60/100.000 in men in Hungary. In the investigators' country the stroke patients are 5-10 years younger as compared to other developed countries. The total stroke mortality in the first 24 months in Hungary is approximately 30%, furthermore 32-42% of the survivors need permanent help in completing their daily routine tasks. Carotid artery disease of atherosclerotic origin is common in the elderly population. The cause of cerebral ischemia in approximately half of the patients is due to the rupture of atherosclerotic plaque with subsequent embolization of thrombus and/or plaque material in the cerebral circulation. Prevention of cerebral ischemia is the goal of pharmacological or surgical treatment. The decision for surgical treatment such as carotid endarterectomy (CEA) or carotid artery stenting (CAS) is based on the degree of stenosis, but incorporating non-invasive measures of plaque composition is expected to improve the selection of patients that will benefit from surgical intervention. The number of asymptomatic patients with carotid stenosis needed to treat to prevent one stroke with endarterectomy is 20, which is quite high compared to 8 in the symptomatic patient group. There is a clear need to identify asymptomatic individuals at high risk of developing future ischemic events to avoid unnecessary surgery. It has been remarked, that the recent AHA (American Heart Association) guideline on the management of significant asymptomatic carotid stenosis recommends that surgery may be considered in highly selected patients. However, no guidance was provided as to which patient is the "highly selected" one.

As of today, no suitable predictive method is available to properly estimate stroke risk in patients with carotid artery stenosis. Carotid artery stenosis is one of the proven risk factors of stroke incidence, but the indication of its intervention is merely the grade of stenosis itself. The current international guidelines suggest intervention for asymptomatic patients only with potentially high risk plaques, but pharmacological treatment is advised for low risk patients. Unfortunately there is no proven and widely accepted system to distinguish these two categories of patients with carotid artery stenosis.

Aims:

The investigators' aim is to establish a stroke risk prediction score system -based on CTA and US plaque morphology and blood sample biomarkers- for asymptomatic carotid artery stenosis patients. A more specific and more accurate system -than the currently applied stroke risk score systems- would allow for the selection of the potentially high risk plaques in asymptomatic patients with borderline grade stenosis.These patients would benefit more from surgical treatment while asymptomatic patients with low risk plaques could avoid the risk of an invasive treatment.

1. Morphological features related to surgical related cerebrovascular events: The investigators plan to overview the clinical records retrospectively to find morphological, hemodynamical and clinical predictors of intra- and early postoperative cause of the cerebrovascular events. An isolated middle cerebral artery carries higher risk of immediate neurological event after carotid endarterectomy with cross-clamping without shunt protection. This project's secondary aims are the following: to compare the accuracy of the CTA and MR imaging in the assessment of the Circle of Willis (CoW) morphology in all patients before CEA and to evaluate changes in CoW morphology before and after CEA, to compare ischemic changes before and after CEA regarding CoW morphology, shunt usage and to evaluate the impact of contralateral carotid occlusion on immediate neurological event (INE) regarding CoW and other supra-aortic morphology. Retrospective assessment of the correlation between intracranial vascular morphology with CTA and intraoperative stroke risk would provide help in perioperative stroke risk prediction and planning of optimal surgical technique.
2. Micro-embolization and carotid plaque analysis: The investigators aim is to define a group of patients in the study cohort, who are clinically asymptomatic, but suffered silent brain ischemia (SBI) before surgery, and to analyze their plaque using a dedicated software for plaque assessment (Medis QAngioCT) and compare to asymptomatic without SBI and symptomatic patients plaques. In Hungary the gold standard of the preoperative imaging of carotid artery stenosis in asymptomatic and symptomatic patients is CTA. These images can be used for plaque analysis that is to identify vulnerable plaque morphology in coronary arteries. The identification of preoperative plaque vulnerability based on the comparison of the ultrasound plaque elastography and contrast enhanced plaque analysis, the transcranial Doppler ultrasound (which can detect microembolisation), cranial DWI-MR for verification of silent recent ischaemic lesions and the histopathology of surgically removed plaques with CTA and US based plaque morphology can define vulnerable plaques related to adverse events.
3. Evaluation of retinal perfusion changes following carotid interventions using OCT angiography in patients with carotid stenosis to assess the influence of carotid stenting and carotid endarterectomy on retinal perfusion using OCTA in patients with significant carotid artery stenosis. Furthermore, this study evaluates the predictive accuracy of retinal microvasculature alterations on the development of postoperative stroke. Carotid artery occlusive disease may result in different vision threatening ocular manifestations, for instance, retinal vascular occlusions and ocular ischemic syndrome (OIS). The diagnosis of carotid stenosis is critical as it is an important risk factor of serious cerebrovascular disease. OCT angiography could be a useful non-invasive method for early diagnosis of patients with carotid stenosis and to evaluate the outcome of carotid interventions. Better identification of patients with carotid stenosis is crucial for the prevention of vision loss and stroke.

ELIGIBILITY:
Inclusion Criteria:

* signed informed consent,
* significant carotid artery stenosis

Exclusion Criteria:

* Age under 50 years
* Neurological event 15 days before operation
* Chronic kidney disease
* Pacemaker or ICD implantation
* Atrial fibrillation

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2019-02-06 (Actual); Primary Completion 2020-11-30 (Estimated); Study Completion 2022-11-30 (Estimated)

PRIMARY OUTCOMES:
Neurological event | Periprocedural (0-78h after the carotid endarterectomy)
  Neurological event can be definitive stroke or transient ischemic attack (TIA). Any neurological events, which can occur in the postoperative 0-78 hours is defined as neurological event. The patients with neurological event will be scored in Rankin scale and will undergo cranial CT and CTA to verify the acute brain ischemia. Patients without any neurological event, who has silent new DWI lesions in postoperative cranial MR, count to be asymptomatic and do not fulfill the positive outcome criteria. Patients with peripheral nerve damage (common complication of cervical operations) count to be asymptomatic and do not fulfill the positive outcome criteria.

CONTACTS AND LOCATIONS:
Overall Officials: Péter Sótonyi, MD PhD, Study Director — Semmelweis University Heart and Vascular Centre
Locations (1):
- Semmelweis University Heart and Vascular Centre, Budapest, Budapest XII, Hungary

IPD SHARING:
Plan to Share IPD: Undecided